CLINICAL TRIAL: NCT02805361
Title: Real World Assessment of Clinical Outcome Changes -Including Month of Ramadan- for Dapagliflozin in Management of Type 2 Diabetes Mellitus
Brief Title: Real World Assessment of Clinical Outcome Changes -Including Month of Ramadan-for Dapagliflozin in Management of Type II Diabetes Mellitus
Acronym: REWARD
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1690R00028
Record Dates: First submitted 2016-06-09; First posted 2016-06-20 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
REWARD is an Non Interventional study aims to describe the changes in the clinical outcomes of Type 2 Diabetes Mellitus patients who are treated with Dapagliflozin for a period of one year including the fasting period of Ramadan

DETAILED DESCRIPTION:
REWARD is a multi-center, post-authorization, prospective, open label, non-interventional, real-life, observational, cohort study. The study is to be conducted at 10-15 sites .

Aims to describe the changes in the clinical outcomes over 1 year as follows:

1. Primary Objective:

   To describe the change in HbAlc from baseline as a parameter for blood glucose control.
2. Secondary Objective:

   To describe the changes from baseline in the following parameters:
   * Total body weight.
   * Total cholesterol, LDL-C, non-HDL-C and triglycerides.
   * Systolic and Diastolic Blood Pressures.
3. Other Objective:

   To capture the frequency & incidence of the following reported adverse events :
   * Hypoglycemic episodes.
   * Volume Depletion.
   * Genital infections.
   * Urinary tract infections.
4. Exploratory Objective:

To describe the combined effect of the hot climate season and fasting Ramadan on the level of total ketone bodies levels in T2DM subjects treated with Dapagliflozin.Description of outcome variables in relation to objectives and hypotheses

ELIGIBILITY:
Inclusion Criteria:

The target population will be selected according to the following inclusion criteria:

* Males and females participants aged 18 years and older who are diagnosed type 2 Diabetic patients- (Based on American Diabetes Association diagnostic criteria (ADA), The ADA defines diabetes as a fasting blood glucose (FBG) of ≥ 126mg/dL or a 2-hour glucose level post oral glucose tolerance test (OGTT) of ≥ 200 mg/dL or HbAJC of ≥ 6.5%).
* Patients treated with Dapagliflozin (as per routine care and in compliance with the locally approved prescribing information) for ≥ 4 weeks and ≤ 16 weeks prior to the recruitment date.
* Patients with CrCl > 60 ml/min or eGFR > 60 ml/min/1.73 m2 should be included in trial.
* Patients providing written informed consent.

Exclusion Criteria:

* Patients with contraindications to Dapagliflozin as per the locally approved prescribing information will be excluded from the study.
* If participating in any clinical trial, the subject cannot take part in this study.
* Patients with clinically significant renal, hepatic, haematological, oncological, endocrine, psychiatric or rheumatic disease.
* Patients who don't have a disease with life expectancy under 1 year.
* Patients with CrCl < 60 ml/min or eGFR < 60 ml/min/1.73 m2 should be excluded from the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females participants aged 18 years and older who are diagnosed type 2 Diabetic patients (Based on American Diabetes Association diagnostic criteria (ADA))
Sampling Method: Non-Probability Sample
Enrollment: 511 (Actual)
Dates: Start 2016-08-21 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
The mean change in HbAlc from mean baseline and at Month 12. | 12 Months
  Primary Variable: To describe the change in HbAlc from baseline as a parameter for blood glucose controL

SECONDARY OUTCOMES:
Changes from baseline in Total body weight | 12 Months
  The mean changes from mean baselines and at Month12 in Total body weight.
Changes from baseline in Total cholesterol | 12 Months
  The mean changes from mean baselines and at Month12 in Total cholesterol.
Changes from baseline in Systolic Blood Pressures | 12 Months
  The mean changes from mean baselines and at Month12 in Systolic Blood Pressures
Changes from baseline in LDL-C | 12 Months
  The mean changes from mean baselines and at Month12 in LDL-C
Changes from baseline in non-HDL-C | 12 Months
  The mean changes from mean baselines and at Month12 in non-HDL-C
Changes from baseline in triglycerides. | 12 Months
  The mean changes from mean baselines and at Month12 in triglycerides
Changes from baseline in Diastolic Blood Pressures | 12 Months
  The mean changes from mean baselines and at Month12 in Diastolic Blood Pressures.

OTHER OUTCOMES:
The frequency & incidence of Hypoglycemic episodes | 12 Months
  The frequency & incidence of the following reported adverse events during the 12 Months period of the study: Hypoglycemic episodes.
The frequency & incidence of Volume Depletion. | 12 Months
  The frequency & incidence of the following reported adverse events during the 12 Months period of the study: Volume Depletion.
The frequency & incidence of Genital infections | 12 Months
  The frequency & incidence of the following reported adverse events during the 12 Months period of the study: Genital infections
Capture influence of the combined effect of fasting and hot climate on the level of total ketone bodies levels in T2DM subjects treated with Dapagliflozin | 12 Months
  Quantitative estimation of capillary ketone bodies will be carried out within 3-months prior Ramadan in selected centers where this is a routine clinic practice. In patients where quantitative estimation of capillary ketone bodies was measured prior to Ramadan, another measurement will be carried out during Ramadan if the date of patient routine follow-up visit coincided with the month of Ramadan. In case visit coincides with only a couple of days of fasting, measurements would be taken into the middle and/or the end of Ramadan. In case someone is recruited during Ramadan, baseline recorded measurements must be prior to Ramadan

CONTACTS AND LOCATIONS:
Overall Officials: Tarek M. Fiad, MBBCH MD FRCPI FRCP, Principal Investigator — Endocrinology Division Departemnt of Medicine, SKMC-UAE
Locations (4):
- Research Site, Kuwait City, Kuwait
- United Arab Emirates (3):
  - Research Site, Abu Dhabi
  - Research Site, Ajman
  - Research Site, Dubai

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1690R00028&attachmentIdentifier=afbae225-295f-40d2-a1e2-54a9e57c3666&fileName=REWARD_STUDY_REPORT_SYNOPSIS_CTT.pdf&versionIdentifier=